CLINICAL TRIAL: NCT02744456
Title: A Pilot Study of N-of-1 Trials of Blood Pressure Medications in Adults With Hypertension
Brief Title: N-of-1 Trials for Blood Pressure Medications in Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Ian Kronish, Associate Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAN9419
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Hypertension; High Blood Pressure
Keywords: Hydrochlorothiazide tablet; Norvasc; Cozaar; amlodipine besylate tablets; losartan potassium tablets; Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Losartan; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N-of-1 trial (Other): Patients with hypertension who are taking none or one BP medication will be will be provided with prescriptions for up to 3 BP medications representative of different BP medication classes (i.e., losartan, an angiotensin system blocking agent; amlodipine, a calcium channel blocker; and hydrochlorothiazide, a thiazide diuretic). Patients will be asked to take each medication for 2 weeks at a low dose, 2 weeks at a medium dose, and then 2 weeks at a high dose; provide health information and identify which medication they prefer to remain on following the N-of-1 trial (i.e., for long-term use).
  Interventions: Drug: Losartan; Drug: Amlodipine; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Losartan — An angiotensin II receptor antagonist drug used mainly to treat high blood pressure.
  Other Names: Losartan potassium tablets; Cozaar
Drug: Amlodipine — A calcium channel blocker and may be used alone or in combination with other antihypertensive and antianginal agents for the treatment of hypertension.
  Other Names: Amlodipine besylate tablets; Norvasc
Drug: Hydrochlorothiazide — A diuretic medication often used to treat high blood pressure and swelling due to fluid build up.
  Other Names: HCTZ; Hydrochlorothiazide tablets

SUMMARY:
Many patients want to know which blood pressure medication is the best for them. In this study, we will test the feasibility of a new approach to determining the best blood pressure medication for individual patients by performing an N-of-1 trial in which patients will have the opportunity to test a series of 3 blood pressure medications at escalating doses while carefully measuring their blood pressure and side-effects. At the end of each of these N-of-1 trials, we will ask patients to complete a questionnaire in which they rate their level of satisfaction with this approach to learning about which is the best blood pressure medication for them.

DETAILED DESCRIPTION:
The goal of this research is to empower hypertensive patients to learn which blood pressure (BP) medication is best for them. Although lifestyle factors such as diet and exercise play an important role, medications may still needed to achieve BP control. Yet, there are substantial differences in the way BP medications affect patients; medications well-tolerated in some, cause severe side-effects in others. Similarly, medications that cause larger reductions in BP in some patients have smaller BP lowering effects in others. Despite this heterogeneity in treatment effects, there are no proven real-world methods to help patients identify the medication most suited to their needs.

One potential approach to individualizing BP treatment decisions is to conduct N-of-1 trials: a multiple crossover design conducted in a single patient. Despite the appeal of this approach, there are few published reports of BP medication N-of-1 trials. Therefore, the objective of this study is to determine the feasibility of conducting an N-of-1 BP medication trial in hypertensive patients. Patients who meet all the eligibility criteria will be asked to monitor their blood pressure and side-effects while taking a series of commonly prescribed blood pressure medications. If they are already taking a blood pressure medication, they will begin by tracking their blood pressure and side-effects while taking this medication for 1 week. They will then be asked to track their blood pressure and side-effects while taking a series of up to three other blood pressure medications (losartan - a renin-angiotensin system blocking agent, amlodipine - a calcium channel blocker, and hydrochlorothiazide - a thiazide diuretic). Each of these medications will be taken for 2 weeks at a time. The specific choice of medications and medication doses will be selected by the study physician. Unless patients have side-effects that lead them to discontinue a medication early, patients will be expected to take each medication at least twice in a balanced sequence (e.g., losartan - amlodipine - HCTZ - HCTZ - amlodipine - losartan). Patients will measure their blood pressure and medication side-effects during the 2nd week on each of these medications. Patients will have the option of escalating or decreasing dosages to identify the single medication/medication dose that best lowers their blood pressure with the least side-effects. Blood pressure will be measured using an Omron home blood pressure monitor. Side-effects will be tracked using a daily e-mailed survey that is completed over the Internet.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 80 years.
* History of physician-diagnosed hypertension.
* Currently not treated with antihypertensive medication but with consensus (from patient and his/her physician; patients with elevated ABPM who are not on treatment will be considered eligible irrespective of office BP if the patient's physician is in agreement with a trial of BP medications) that antihypertensive medication should be initiated; or being treated with one antihypertensive medication.
* No history of suspected or confirmed white coat hypertension (elevated clinic BP but non-elevated out-of-clinic BP either by home BP monitoring or ABPM).
* Easy access to and regular use of e-mail as they will need to be able to respond to Qualtrics surveys at regular intervals during the self-monitoring period.
* Established relationship with an accessible primary care provider.
* Primary care provider gives permission to participation in an N-of-1 trial.

Exclusion Criteria:

* Severe hypertension (office BP = 180/110 mm Hg).
* History of myocardial infarction, heart failure, atrial fibrillation, or chronic kidney disease as these patients have guideline recommended indications for specific classes of BP medications.
* Electrolyte abnormality; if no electrolyte panel is available in the prior 6 months, then one will be ordered for purposes of the study.
* Known drug allergy or intolerance to angiotensin receptor blocker, calcium channel blocker, or thiazide diuretic.
* Prescribed BP medication for indication other than hypertension (e.g., migraine headache prophylaxis, enlarged prostate).
* Primary care provider permission not obtained.
* Non-English speaking.
* No regular (daily) access and use of e-mail as participants will need to be able to respond to emailed links to surveys for completion of self-monitoring symptoms.
* Unable to provide informed consent or adhere to study protocol due to cognitive impairment, mental illness, or other reasons.
* Unable to monitor BP at home using an automatic BP machine due to physical or mental impairments.
* Unable to track side effects of medications due to physical or mental impairments including literacy problems.
* Arm circumference <9 inches or >17 inches as these sizes do not accommodate the range of BP cuff sizes that are available for the automatic BP machine.
* Unavailable for follow-up during the study period due to severe medical illness or other reasons.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Participants satisfied with participating in N-of-1 trial | 4 months
  Question assessing helpfulness of participating in N-of-1 trial methodology with respecting to managing their hypertension

SECONDARY OUTCOMES:
Participants satisfied with blood pressure regimen | 5 months (or 1 month after completing N-of-1 trial)
  Treatment Satisfaction Questionnaire for Medication

OTHER OUTCOMES:
Adherence to antihypertensive medication | 5 months (or 1 month after completing N-of-1 trial)
  Voils Nonadherence Measure

CONTACTS AND LOCATIONS:
Overall Officials: Ian Kronish, MD, MPH, Principal Investigator — Columbia Univeristy Medical Center
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD is currently presented in the manuscript due to the N-of-1 study design. Participant consent forms will be reviewed with the Columbia University IRB to determine whether we have permission to share de-identified IPD with other researchers.

REFERENCES:
- [Derived] Kronish IM, Cheung YK, Shimbo D, Julian J, Gallagher B, Parsons F, Davidson KW. Increasing the Precision of Hypertension Treatment Through Personalized Trials: a Pilot Study. J Gen Intern Med. 2019 Jun;34(6):839-845. doi: 10.1007/s11606-019-04831-z. Epub 2019 Mar 11. PMID 30859504